CLINICAL TRIAL: NCT00109798
Title: Phase II Trial of Salvage Chemotherapy With Temozolomide in Combination With Topotecan for Primary CNS Lymphoma
Brief Title: Temozolomide and Topotecan in Treating Patients With Primary CNS Lymphoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sub-Investigator reloacted to another institution
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCM IRB#H-16155; CDR0000427313 (Other: Principal Investigator)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Central Nervous System Tumors; Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma | interventions — Temozolomide; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide, Topotecan (Experimental): Patient will take on days 1-5 of a 28-days schedule. Take Topotecan on days 2-6 of the 28 day schedule
  Interventions: Drug: temozolomide; Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: temozolomide — Patient will take drug on day 1-5 of 28 day schedule
  Other Names: Temodar
Drug: topotecan hydrochloride — Patient will have IV on days 2-6 on a 28-day schedule
  Other Names: Topotecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide and topotecan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving temozolomide together with topotecan works in treating patients with primary CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete radiologic response rate in patients with primary CNS lymphoma treated with salvage chemotherapy comprising temozolomide and topotecan.

Secondary

* Determine the median and failure-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the overall response rate in patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive oral temozolomide once daily on days 1-5 and topotecan IV over 30 minutes once daily on days 2-6. Treatment repeats every 28 days for 6-8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 6-25 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

DISEASE CHARACTERISTICS:

* Histologically confirmed primary CNS lymphoma at initial diagnosis
* Measurable tumor by radiography
* Failed* OR is not a candidate for first-line high-dose systemic methotrexate-based chemotherapy with or without radiotherapy NOTE: *Failure is defined as relapse, progression, or failure to achieve a complete response

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 50-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL

Hepatic

* SGOT and SGPT ≤ 3 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine clearance > 40 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No known allergy to temozolomide or topotecan
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or stage I or II cancer in complete remission
* No other major medical illness or psychiatric impairment that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic growth factors

Chemotherapy

* See Disease Characteristics
* At least 6 weeks since prior nitrosoureas
* At least 2 weeks since prior methotrexate

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Other

* Recovered from all prior therapy
* At least 4 weeks since prior non-nitrosourea cytotoxic drugs (except methotrexate)
* At least 4 weeks since prior systemic investigational agents
* At least 2 weeks since prior non-cytotoxic antitumor drugs
* No other concurrent antitumor therapy

EXCLUSION CRITERA

1. Patients who are pregnant or breastfeeding, or females of childbearing potential not using adequate contraception.
2. Known allergy to temozolomide or topotecan.
3. Severe vomiting or other inability to administer medications orally.
4. Major medical illnesses or psychiatric impairment that in the investigator's opinion will prevent administration or completion of the protocol therapy and/or will interfere with follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Rate of complete radiologic response (CR) | July 2006

SECONDARY OUTCOMES:
Median overall survival | July 2006
Failure-free survival | July 2006
Toxicity | July 2006
Overall response rate (CR and partial response) | July 2006

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Z. New, MD, Study Chair — Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: No